CLINICAL TRIAL: NCT00865696
Title: A Relative Bioavailability Study of 15 mg Mirtazapine Tablets Under Fasting Conditions
Brief Title: A Relative Bioavailability Study of Mirtazapine 15 mg Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Meena Venugopal, Director, Clinical R&D, Actavis Inc
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: R00-435
Record Dates: First submitted 2009-03-17; First posted 2009-03-19 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Mirtazapine; Healthy subjects
MeSH Terms: interventions — Mirtazapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Mirtazapine 15 mg tablets, single dose
  Interventions: Drug: Mirtazapine 15 mg tablets, single dose
- B (Active Comparator): REMERON® 15 mg tablets, single dose
  Interventions: Drug: REMERON® 15 mg tablets, single dose

INTERVENTIONS:
Drug: Mirtazapine 15 mg tablets, single dose — A: Experimental Subjects received Purepac formulated products under fasting conditions
  Other Names: Mirtazapine
  Arms: A
Drug: REMERON® 15 mg tablets, single dose — B: Active comparator Subjects received Organon Inc. formulated products under fasting conditions
  Other Names: Mirtazapine
  Arms: B

SUMMARY:
The purpose of this study is to compare the relative bioavailability of 15 mg Mirtazapine Tablets by Purepac Pharmaceutical Co with that of 15 mg REMERON® Tablets by Organon Inc. following a single oral dose (1 x 15 mg) in healthy adult volunteers under fasting conditions.

DETAILED DESCRIPTION:
Study Type: Interventional Study Design: Randomized, single dose, two-way crossover study under fasting conditions

Official Title: A Relative Bioavailability of 15 mg Mirtazapine Tablets Under Fasting Conditions

Further study details as provided by Actavis Elizabeth LLC:

Primary Outcome Measures:

Rate and Extend of Absorption

ELIGIBILITY:
Inclusion Criteria:

* Screening Demographics: All volunteers selected for this study will be healthy men and women 18 years of age or older at the time of dosing. The weight range will not exceed ± 20% for height and body frame as per Desirable Weights for Men -1983 Metropolitan Height and Weight Table or as per Desirable Weights for Women - 1983 Metropolitan Height and Weight Table.
* Screening Procedures: Each volunteer will complete the screening process within 30 days prior to Period I dosing. Consent documents for both the screening evaluation and HIV antibody determination will be reviewed, discussed, and signed by each potential participant before full implementation of screening procedures.
* Screening will include general observations, physical examination, demographics, medical and medication history, an electrocardiogram, sitting blood pressure and heart rate, respiratory rate and temperature. -The physical examination will include, but may not be limited to, an evaluation of the cardiovascular, gastrointestinal, respiratory and central nervous systems.
* The screening clinical laboratory procedures will include:

  * HEMATOLOGY: hematocrit, hemoglobin, WBC count with differential; RBC count, platelet count
  * CLINICAL CHEMISTRY: serum creatinine, BUN, glucose, AST(GOT), ALT(GPT), albumin, total bilirubin, total protein, and alkaline phosphatase;
  * HIV antibody and hepatitis B surface antigen screens;
  * URINALYSIS: by dipstick, microscopic examination if dipstick positive; and .
  * URINE DRUG SCREEN: ethyl alcohol, amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine metabolites, opiates and phencyclidine.
  * SERUM PREGNANCY SCREEN (female volunteers only)
* If female and:

  * of childbearing potential, is practicing an acceptable barrier method of birth control for the duration of the study as judged by the investigator(s), such as condoms, sponge, foams, jellies, diaphragm; intrauterine device (IUD), or abstinence
  * is postmenopausal for at least I year; or
  * is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy)

Exclusion Criteria:

* Volunteers with a recent history of drug or alcohol addiction or abuse.
* Volunteers with the presence of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease (as determined by the medical investigator).
* Volunteers whose clinical laboratory test values are outside the accepted reference range and when confirmed on re-examination are deemed to be clinically significant.
* Volunteers demonstrating a positive hepatitis B surface antigen screen or a reactive HIV antibody screen.
* Volunteers demonstrating a positive drug abuse screen when screened for this study.
* Female volunteers demonstrating a positive pregnancy screen.
* Female volunteers who are currently breastfeeding.
* Volunteers with a history of allergic response(s) to mirtazapine or related drugs.
* Volunteers with a history of clinically significant allergies including drug allergies.
* Volunteers with a clinically significant illness during the 4 weeks prior to Period I dosing (as determined by the medical investigator).
* Volunteers who currently use tobacco products.
* Volunteers who have taken any drug known to induce or inhibit hepatic• drug metabolism in the 30 days prior to Period I dosing.
* Volunteers who report donating greater than 150 mL of blood within 30 days prior to Period I dosing. All subjects will be advised not to donate blood for - Volunteers who have donated plasma (e.g. plasmapheresis) within 14 days prior to Period I dosing. All subjects will be advised not to donate plasma for four weeks after completing the study.
* Volunteers who report receiving any investigational drug within 30 days prior to Period I dosing.
* Volunteers who report taking any systemic prescription medication in the 14 days prior to Period I dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2001-09; Primary Completion 2001-09 (Actual); Study Completion 2001-09 (Actual)

PRIMARY OUTCOMES:
Rate and Extend of Absorption | 120 hours

CONTACTS AND LOCATIONS:
Overall Officials: James D. Carlson,, Pharm.D,, Principal Investigator — PRACS Institute, Ltd.
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States